CLINICAL TRIAL: NCT05661461
Title: A Phase 1, Open-label, Dose-escalation Study to Assess Safety and Pharmacokinetics of Nab-Sirolimus in Patients With Locally Advanced or Metastatic Solid Tumors and Moderate Liver Impairment
Brief Title: Dose-escalation Study to Assess Safety and Pharmacokinetics of Nab-Sirolimus in Patients With Locally Advanced or Metastatic Solid Tumors and Moderate Liver Impairment
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HEP-001
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Tumor, Solid; Tumor; Advanced Solid Tumor
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): nab-Sirolimus
  Interventions: Drug: nab-sirolimus

INTERVENTIONS:
Drug: nab-sirolimus — This is a phase 1, multi-center, open-label, dose-escalation study of nab-sirolimus in adult patients with locally advanced or metastatic solid tumors and moderate hepatic impairment or normal hepatic function.
  Other Names: ABI-009, nab-rapamycin, albumin-bound rapamycin

SUMMARY:
This is a phase 1, multi-center, open-label, dose-escalation study of nab-sirolimus in adult patients with locally advanced or metastatic solid tumors and moderate hepatic impairment or normal hepatic function.

DETAILED DESCRIPTION:
This is a phase 1, multi-center, open-label, dose-escalation study of nab-sirolimus in adult patients with locally advanced or metastatic solid tumors and moderate hepatic impairment or normal hepatic function. Eligible patients will receive nab-sirolimus by intravenous (IV) infusion over 30 minutes (+10 min) on Days 1 and 8.

ELIGIBILITY:
Inclusion Criteria:

* For All Patients

  1. Willing and able to provide informed consent and comply with protocol requirements for the duration of the study.
  2. Male or female patients at least 18 years of age at the time of signing the informed consent form.
  3. Histologically confirmed locally advanced or metastatic solid tumors that is measurable or non-measurable.
  4. Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
  5. Adequate hematologic counts:

     * Absolute neutrophil count (ANC) ≥1.0 × 109 /L (growth factor support allowed)
     * Platelet count ≥75,000/mm 3 (75 × 10 9 /L) (transfusion and/or growth factor support allowed)
     * Hemoglobin ≥8.0 g/dL (transfusion and/or growth factor support allowed)
  6. Creatinine clearance ≥30 mL/min as assessed by the Cockcroft-Gault equation:

     Creatinine Clearance ≥30 = (140 - age) × (weight[kg] / (72 x SCr[mL/min]_ x 0.85, if female
  7. Fasting serum triglyceride must be ≤300 mg/dL; fasting serum cholesterol must be

     ≤350 mg/dL.
  8. Male or non-pregnant and non-breastfeeding female:

     * Females of child-bearing potential must agree to use highly effective contraception or abstinence without interruption from 28 days prior to first dose throughout 3 months after last dose and have a negative pregnancy test (urine or serum) result at screening and after the end of study treatment. A second form of birth control is required even if she has had a tubal ligation.
     * Male patients must practice abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study and throughout 3 months after last dose. A second form of birth control is required even if he has undergone a successful vasectomy.
  9. Minimum of 4 weeks since major surgery, completion of radiation, or completion of all prior systemic anticancer therapy, or at least 5 half-lives if the prior therapy is a single agent small-molecule therapeutic, and in either case adequately recovered from the acute toxicities of any prior therapy (including neuropathy) to Grade ≤1. For Patients with Normal Hepatic Function
  10. Normal hepatic function (total bilirubin ≤ upper limit of normal [ULN] and aspartate aminotransferase [AST] ≤ULN). For Patients with Moderate Hepatic Impairment
  11. Moderate hepatic impairment (total bilirubin 1.5-3.0 × ULN and any level of AST)

Exclusion Criteria:

1. Received prior treatment with an mTOR inhibitor within 4 weeks prior to first dose.
2. Patients who have any severe and/or uncontrolled medical or psychiatric conditions or other conditions that could affect their participation including:

   1. Patients with meningeal carcinomatosis, leptomeningeal carcinomatosis, spinal cord compression, untreated brain metastases or symptomatic or unstable brain metastases. Note: Patients with stable brain metastases (defined as asymptomatic or no requirement for high-dose [defined as dexamethasone 10 mg daily or higher] or increasing dose of systemic corticosteroids) and without imminent need of radiation therapy are eligible. If applicable, patients must have completed brain radiation therapy and recovered adequately from any associated toxicity and/or complications prior to eligibility assessment. For patients who have received prior radiation therapy, post-treatment magnetic resonance imaging (MRI) scan should show no increase in brain lesion size/volume.
   2. Unstable angina pectoris, symptomatic congestive heart failure (New York Heart Association, NYHA class III or IV), myocardial infarction ≤6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
   3. Pre-existing severely impaired lung function. If a patient has a pre-existing pulmonary condition, eligible patients should have a spirometry and diffusing capacity for carbon monoxide (DLCO) that is >50% of the normal predicted value and/or O2 saturation that is >88% at rest on room air (Note: spirometry and pulmonary function tests [PFTs] not required to be performed unless clinically indicated).
   4. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy. Note, controlled non melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer, or other adequately treated carcinoma-in-situ may be eligible, after documented discussion with the Medical Monitor.
   5. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg).
   6. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
   7. Individuals with known human immunodeficiency virus (HIV) infection are excluded from this study as combination antiretroviral therapy could potentially result in significant pharmacokinetic interactions. In addition, these individuals are at increased risk of serious infections due to the immunosuppressive effects of mTOR inhibition.
   8. Active Hepatitis B or Hepatitis C, with detectable viral load. Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients.
3. Have active severe (Grade ≥3) infection requiring intravenous (IV) antibiotics (contact medical monitor for clarification).
4. High-dose systemic corticosteroids (>10 mg of prednisone or its equivalent) are not permitted within 2 weeks of first dose. However, inhaled, intranasal, intra articular, and topical steroids are allowed.
5. Have a history of Gilbert's disease.
6. Any condition that in the opinion of the Investigator would place the patient at an unacceptable risk or cause the patient to be unlikely to fully participate or comply with study procedures.

   For Patients with Moderate Hepatic Impairment
7. Had a clinical exacerbation of liver disease within the 2-week period prior to first dose (ie, abdominal pain, nausea, vomiting, anorexia, or fever).
8. Have clinically demonstrable, tense ascites.
9. Had evidence of acute viral hepatitis within 1 month prior to first dose.
10. Have evidence of hepatorenal syndrome.
11. Have a transjugular intrahepatic portosystemic shunt.
12. Have active stage 3 or 4 encephalopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
MTD for patients with moderate hepatic impairment | Through Day 22
Maximum concentration (Cmax) | Time 0
Area under the serum concentration-time curve | Time 0 to time of the last quantifiable concentration (AUC 0-last)
Area under the serum concentration-time curve | Time 0 to 168 hours (AUC 0-168)

SECONDARY OUTCOMES:
Area under the serum concentration-time curve | Time 0 extrapolated to infinity (AUC0-inf)
Time to maximum observed serum concentration (T max) | Time 0 to 168 hours (AUC 0-168)
Clearance (CL) | Time 0 to 168 hours (AUC 0-168)
Total volume of distribution during the terminal phase (V z ) | Time 0 to 168 hours (AUC 0-168)
Steady-state volume of distribution (V ss) | Time 0 to 168 hours (AUC 0-168)
Terminal elimination rate constant (λz ) | Time 0 to 168 hours (AUC 0-168)
Terminal elimination half-life (t½ ) | Time 0 to 168 hours (AUC 0-168)
Accumulation ratio based on Cmax | Time 0 to 168 hours (AUC 0-168)
Accumulation ratio based on AUC0-168 | Time 0 to 168 hours (AUC 0-168)
Percent area under the serum concentration-time curve extrapolated (%AUCextrap ) | Time 0 to 168 hours (AUC 0-168)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
  - START Mountain Region, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No